CLINICAL TRIAL: NCT02059772
Title: Evaluation of an Additional Therapeutic Approach to Diabetic Macular Edema by Combining Standard Therapy (Intravitreal Injection of a VEGF-inhibitor) With Micropulse Diode Laser Treatment in a Randomized, Controlled Proof of Concept Study
Brief Title: Combination of Standard Lucentis Therapy With Micropulse Diode Laser for the Treatment of Diabetic Macular Edema
Acronym: ReCaLL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReCaLL-2013
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Experimental): Standard therapy of diabetic macular edema with Lucentis (ranibizumab) according to SmPC
  Interventions: Drug: ranibizumab
- Treatment Group (Experimental): Combination of standard therapy of Lucentis (ranibizumab) according to SmPC and micropulse diode laser treatment
  Interventions: Drug: ranibizumab; Procedure: micropulse diode laser

INTERVENTIONS:
Drug: ranibizumab
  Other Names: Lucentis
Procedure: micropulse diode laser
  Arms: Treatment Group

SUMMARY:
The primary objective of this study is to evaluate if a combination therapy with micropulse diode laser treatment shows non inferiority on visual acuity within 12 months in comparison to standard therapy (intravitreal injection of ranibizumab only).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-ischemic diabetic macular edema with resulting reduction in visual functionality by determination of best corrected visual acuity (BCVA), ophthalmologic investigation, SD-OCT, FAG and anamnesis
* BCVA between 0.05 and 0.6 or retinal thickness > 300 µm determined by SD-OCT
* The informed consent form must be signed before any study specific tests or procedures are done
* Confirmation of the subject's health insurance coverage prior to the first screening visit
* Age at least 18 years (inclusive) at the first screening visit
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Severe ischemic maculopathy of the study eye
* Active neovascularization of iris or retina in the study eye
* History of intravitreal injection of VEGF-inhibitor or steroids in study eye within the last 3 month
* Pathologies of the anterior segment of the study eye with reduced visual acuity (e.g. corneal opacification, advanced cataract)
* Advanced glaucoma with central defects of the visual field in study eye
* Retinal pathologies with reduced visus (e.g. central scars, age related macular degeneration) in study eye
* Retinal vascular occlusion in medical history of study eye
* Active or suspected ocular or periocular infections
* Active intraocular inflammation in study eye
* Intraocular surgery of study eye within the last 6 months
* Laser therapy of study eye within the last 6 months
* Systemic steroid therapy within the last 3 month
* HbA1c >10%
* Systolic blood pressure above 170 mmHg and diastolic blood pressure above 110 mmHg (after at least 3 min in supine position)
* Pregnant or breast-feeding woman and woman without adequate method of contraception.
* Known hypersensitivity to the active substance or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
change in best corrected visual acuity (BCVA) | baseline, 12 month

SECONDARY OUTCOMES:
change in central macular thickness | baseline, 12 month
number of intravitreal Lucentis injections | within 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Klio Ai Becker, MD, Study Chair
Locations (1):
- Klinik für Augenheilkunde, Klinikum Chemnitz gGmbH, Chemnitz, Germany

REFERENCES:
- [Derived] Furashova O, Strassburger P, Becker KA, Engelmann K. Efficacy of combining intravitreal injections of ranibizumab with micropulse diode laser versus intravitreal injections of ranibizumab alone in diabetic macular edema (ReCaLL): a single center, randomised, controlled, non-inferiority clinical trial. BMC Ophthalmol. 2020 Jul 29;20(1):308. doi: 10.1186/s12886-020-01576-w. PMID 32727496